CLINICAL TRIAL: NCT02331719
Title: Minimally Invasive Subcortical Parafascicular Access for Clot Evacuation
Brief Title: Evaluation of Minimally Invasive Subcortical Parafascicular Access for Clot Evacuation
Acronym: MiSPACE
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 14-39E
Record Dates: First submitted 2014-12-17; First posted 2015-01-06 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Hemorrhage
Keywords: intracerebral hemorrhage; subcortical intracerebral hemorrhage; ICH; parafascicular minimally invasive subcortical access
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MiSPACE Eligible Cohort: This will be a prospective record review of patients where the MiSPACE technique is being/was used for the treatment of their ICH.
- Historical Cohort: This is a retrospective records review of patients who received either medical intervention or conventional surgical intervention for the treatment of their ICH.

SUMMARY:
Intracerebral hemorrhage (ICH) is the most severe form of stroke: early mortality is 40%, and 80%-of survivors are physically disabled with high rates of cognitive impairment and depression.

In an effort to address the issues with conventional treatments, a new integrated systematic approach has been developed. This approach utilizes an educational process where specific core competencies (pillars) of mapping, navigation, access, optics and automated resection have been integrated into a single standardized system to deliver targeted therapy for an individual patient based on location and patient factors. This system has demonstrated safety and efficacy in oncology patients and is also FDA approved for use in the ICH patient population as well.

This registry will collect data form multiple site that preform the MiSPACE procedure as part of clinical care. The intent of this registry is to collect data on the economic impact as well as clinical outcomes using the MiSPACE approach with the integrated technology in the early treatment of ICH.

DETAILED DESCRIPTION:
Aurora Health Care is serving as the coordinating center and will prepare Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, and reporting for adverse events.

Sites will identify, recruit, obtain consent for subjects and collect data using standard forms; these activities will be monitored remotely by the coordinating site. Data from the participating hospitals will be checked for heterogeneity, queried and subsequently pooled. Baseline patient characteristics and demographics, Hemphill and Essen predictive scores, NIHSS stroke severity score, functional status from the Barthel index and mRS score, and ICH volumetric assessments, will be presented as means, medians, or proportions, as appropriate. Eligibility and consent rates will be derived for each center.

Analyses will be largely descriptive in nature. Follow-up assessments at 30 and 90 days, for composite outcome of death or disability (defined as mRS>2), and death and disability separately, will be described with proportions. Tallies of surgical complications will also be derived as separate outcomes.

Analysis of 30- and 90-day status will entail an informal comparison for the purposes of providing preliminary evidence and for planning of a larger comparative trial. The proportion of patients under experimental treatment who suffer from death or dependency at 30-days, as determined by cutoffs on the modified Rankin Scale with exact binomial upper and lower 90% confidence limits will be used in a comparison to our criteria of: (1) 65% (historical proportion of patients under medical management, unselected for baseline risk), and (2) 50% (proportion of patients under other minimally invasive surgical techniques unselected for baseline risk). This confidence limit comparative approach provides a flexible method of assessment of non-inferiority, equivalence, and superiority. The unselected population will, however, be a mix of patients at different levels of baseline risk, and so a follow-up stratified analysis will be conducted if counts permit. The unselected population will be matched using demographics, lesion characteristics and comorbidities as close as possible to the study group. A heterogeneity index will be used for comparison. As a corollary to this analysis, baseline predictive scores (translated from scores to percentages/risks) will be used to calculate expected counts of 30 and 90 day status stratified within the 0-3 range of the Hemphill ICH score and 0-10 range of the Essen ICH score, and these expected counts will be compared to observed counts using a Fisher Exact Test.

Fifty (50) patients were chosen as a convenient sample size, based on enrollments from all of the participating hospitals, with recruitment accomplished in a reasonable timeframe of 2 years. About 65% of unselected patients with ICH (that is, not stratified by baseline predicted risk) have a documented 30- day composite outcome of death or dependency under medical management. Reviews of other types of minimallyinvasive ICH surgeries provide evidence of significantly improved outcomes (meta-analysis odds ratio 0.54 (0.39, 0.76)). An odds ratio of 0.54 indicates a reduction in risk from 65% to about 50% (15% absolute reduction).

Assuming the new procedure is truly at least as effective as other minimally invasive surgeries (50% 30-day composite outcome risk), and therefore 15% more effective than conventional management, 50 patients provides 66% surity that a 95% 1-sided confidence interval will exclude the chance that the new procedure is worse than medical management.

An alternative method of framing this, based on an exact one-sided binomial test of a one-sample proportion and an alpha level of 5%, is that a sample size of 50 patients provides approximately 66% surity/power that the new procedure is superior to medical management (i.e., lower than 65% suffering from death or poor functional outcomes). The computed critical value for this test, to provide some initial evidence of superiority, is observing no more than 26 patients (out of 50) suffering from death or dependency under the new surgical procedure. The surity/power of 66% used as an assumption above is permissive. The study size and preliminary nature of the results will not be sufficient to perform robust statistical testing for superiority or non-inferiority of the new parafascicular ICH-evacuation technique, though results from this registry will provide a crucial first look at effectiveness, and health costs.

ELIGIBILITY:
Inclusion Criteria:

* Presented with acute symptomatic supratentorial primary ICH diagnosed by CT
* Has made the clinical treatment decision to have parafascicular minimally invasive subcortical (MIS) access to treat subcortical intracerebral hemorrhage (ICH) using the systems approach outlined in this protocol
* 18 - 80 years old
* Symptom onset to surgery < 24 hours (target < 8hours)
* Presurgical Glascow Coma Score ≥ 8
* Hematoma volume < 60ml
* Minimal or no ventricular extension (corresponding to 50% or less of each ventricle)

Exclusion Criteria:

* Suspected secondary ICH
* Infratentorial ICH
* Isolated IVH
* Uncorrected coagulopathy
* Significant premorbid disability (mRS>1)
* Hydrocephalus
* Contraindication to safe surgical procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for subcortical intracerebral hemorrhage (ICH) using a systems approach which integrates five separate core competencies for safe and consistent parafascicular minimally invasive subcortical (MIS) access
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Overall surgical performance. | 30 days after procedure
  Overall surgical performance is a composite outcome measure that will be assessed by evaluating a number of events and outcomes. Data will be collected on any surgical complications (defined as peri-operative blood loss, thrombotic events, infections, neurological worsening, seizures, metabolic disturbances, and cardiopulmonary events, within 30 days of surgery). Data from re-admissions within the first 30 days will also be included. In addition, data regarding the duration of surgery, time to reach the hematoma, intra-operative monitoring, blood transfusion, use of hemostatic agents, use of post-operative ICP monitoring, residual post-operative hematoma volumes, and post-operative recurrence of hematoma will also be collected.

SECONDARY OUTCOMES:
Peri-operative complications following parafascicular ICH evacuation. | 90 days after procedure
  Peri-operative complications following parafascicular ICH evacuation will be described and quantified.
  Data will be collected on any surgical complications (defined as peri-operative blood loss, thrombotic events, infections, neurological worsening, seizures, metabolic disturbances, and cardiopulmonary events, within 30/90 days of surgery).
30-day clinical outcomes of patients who had parafascicular ICH-evacuation surgery | 30 days after procedure
  A mRS-certified investigator/delegate will perform a clinical assessment at 30-days and 90-days. In cases where a subject is discharged and unable to attend a follow-up appointment, a standardized telephone mRS interview will be conducted.
90-day clinical outcomes of patients who had parafascicular ICH-evacuation surgery | 90 days after procedure
  A mRS-certified investigator/delegate will perform a clinical assessment at 30-days and 90-days. In cases where a subject is discharged and unable to attend a follow-up appointment, a standardized telephone mRS interview will be conducted.
Inpatient care costs of patients undergoing Parafascicular ICH surgery and patients managed with medical treatment alone or those with conventional surgical treatment. | 90 days after procedure
  An economic analysis comparing inpatient care costs of patients undergoing Parafascicular ICH surgery to patients managed with medical treatment alone or those with conventional surgical treatment. will be completed.
  We will present all the financial results in a relative form using the costreimbursement ratio (CRR); the CRR is simply the ratio of the total cost per patient to the total reimbursement per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Amin B Kassam, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (8):
- United States (8):
  - University Of Arkansas of Medical Sciences, Little Rock, Arkansas
  - University of Colorado, Aurora, Colorado
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - IU Health Neuroscience Center, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Riverside Methodist Hospital (OhioHealth), Columbus, Ohio
  - Aurora Health Care, Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No